CLINICAL TRIAL: NCT06067087
Title: Prognostic Understanding in Patients Receiving Enhanced Supportive Care (ProgESC Study)
Brief Title: Prognostic Understanding in ESC (ProgESC Study)
Status: Completed | Type: Observational
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Other Study IDs: EDGE 158645; IRAS 328196 (Other: Integrated Research Application System)
Record Dates: First submitted 2023-09-27; First posted 2023-10-04 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2025-01

CONDITIONS: Advanced Cancer
Keywords: Prognostic understanding; Enhanced Supportive Care Team; Quality of life; Anxiety; Depression; Satisfaction
MeSH Terms: conditions — Anxiety Disorders; Depression; Personal Satisfaction

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with advanced cancer: Patients with advanced cancer that are referred to the Enhanced Supportive Care Team at University College London Hospital

SUMMARY:
This study aims to assess how aware patients with advanced cancer are about their prognosis when they are referred to an Enhanced Supportive Care (ESC) service. Further, the study aim to assess the relationship between patients prognostic understanding and their mental health, quality of life, trust in medical professionals as well as their perception of the care they receive.

The study will involve adult patients with advanced cancer who are referred to the ESC service at London University College Hospital. Patients who agree to participate will provide consent and answer a questionnaire. The questionnaire will cover their prognostic awareness, psychological symptoms, and quality of life. It takes about 20 minutes to complete and can be done online via RedCap

DETAILED DESCRIPTION:
Background:

Prognostic awareness among patients with life-limiting diseases has been shown to be associated with less depression, better quality of care and earlier referral to palliative care. Moreover, accurate understanding of their illness may support patients to make informed decisions about their future in alignment with their preferences, values or needs.

Supportive care in cancer is the prevention and management of the adverse effects of cancer and its treatment. This includes management of physical and psychological symptoms and side effects. Enhanced Supportive Care (ESC) is a relatively new initiative implementing early supportive care in patients with advanced cancer.

Although studies have shown that a large proportion of patients with advanced cancer remain unaware that their disease is not curable, research regarding prognostic awareness in patients referred to Enhanced Supportive Care (ESC) services is still scarce.

A deeper knowledge of the factors and patient characteristics associated with prognostic awareness is an important first step to develop interventions to improve prognostic communication and thereby to facilitate delivery of high-quality ESC.

General aim:

The ESC team at University College London Hospital is embedded within the oncology outpatient service, providing specialist symptom control and Advanced Care Planning to patients with advanced cancer.

The primary aim of this study is to better understand the prognostic awareness of patients referred to the ESC service. A secondary aim is to evaluate the relationship between patients' prognostic awareness and levels of psychological distress, quality of life, trust in medical professionals and perceived quality of care.

Patient population:

Consecutive adult patients with advanced cancer referred to the ESC service will be eligible to participate. Patients unable to complete questionnaires due to cognitive impairment such as dementia will be excluded. Patients who have already been referred to community palliative care services will also be excluded.

Methods:

This will be a cross-sectional prospective study. Potentially eligible patients will be identified by members of the ESC team and will be informed about the study. Interested patients will then discuss the study with the research team and will be invited to participate. After informed consent has been obtained, participants will complete a questionnaire which will cover their level of prognostic awareness, psychological symptoms, and quality of life). The questionnaire will take approximately 20 minutes to complete. The questionnaire can be completed online via RedCap.

Endpoints:

The primary endpoint of this study is the level of patients' prognostic awareness, which will be assessed by the Prognosis and Treatment Perception Questionnaire. This questionnaire has previously been successfully used in research to assess patients' information preferences, perceptions about their prognosis and the goals of therapy and communication preferences about end-of-life care.

Secondary endpoints will be (a) patients' preferences for receiving prognostic information assessed through the Prognosis and Treatment Perception Questionnaire (b) symptoms of depression evaluated through the Patient Health Questionnaire-2 (PHQ-2), (c) symptoms of anxiety evaluated through the Generalized Anxiety Disorder 2-item (GAD-2), (d) quality of life and (d) patients' trust in their medical team and (e) other aspects of perceived quality of care, rated on a visual analogue scale (NRS) from 0-10.

Sample size and statistics:

The investigators will conduct univariable and multivariable regression analyses to evaluate associations between sociodemographic or clinical variables and outcomes. The investigators aim to include 100 patients. This will give us at least 10 degrees of freedom to assess association of potential risk factors with outcome and to evaluate confounders in a multivariable analysis.

Discussion: This will be the first prospective study to assess prognostic awareness among cancer patients referred to ESC services in a British setting. Identifying covariates for prognostic unawareness and psychological burden among patients with advanced cancer will inform the future development of strategies to improve care and communication with this patient group.

ELIGIBILITY:
Inclusion Criteria:

* All participants aged 18 and older with advanced cancer referred to the ESC team will be eligible for this study.

Exclusion Criteria:

* Younger than 18 years
* Insufficient English language to complete questionnaires
* cognitive impairment
* Participants who, in the opinion of the member of the ESC team, would not be appropriate to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Population: Consecutive patients with advanced cancer being referred to the Enhanced Supportive Care Team
  Setting: UCH Macmillan Cancer Centre
Sampling Method: Non-Probability Sample
Enrollment: 91 (Actual)
Dates: Start 2023-11-15 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2024-08-31 (Actual)

PRIMARY OUTCOMES:
Patients' prognostic understanding | within 1 week after patient assessment by the Enhanced Supportive Care Team
  Patients' prognostic understanding about their illness assessed through the Prognosis and Treatment Perception Questionnaire. This questionnaire assesses patient beliefs regarding the likelihood of cure, the preference for receiving prognostic information as well as the perceived helpfulness of knowing about prognosis

SECONDARY OUTCOMES:
Perceived value of prognostic information | within 1 week after patient assessment by the Enhanced Supportive Care Team
  Assessed through the Prognosis and Treatment Perception Questionnaire. This questionnaire assesses patient beliefs regarding the likelihood of cure, the preference for receiving prognostic information as well as the perceived helpfulness of knowing about prognosis

OTHER OUTCOMES:
Symptoms of anxiety | within 1 week after patient assessment by the Enhanced Supportive Care Team
  Patients' symptoms of anxiety assessed through the Generalized Anxiety Disorder 2-item. This scale has a range from 0 to 6 points with higher scores indicating more symptoms of anxiety. A score of 3 points is considered a cut-off point, in which further evaluation is recommended.
Symptoms of depression | within 1 week after patient assessment by the Enhanced Supportive Care Team
  Patients' symptoms of depression assessed through the Patient Health Questionnaire-2. This scale has a range from 0 to 6 points with higher scores indicating more depressive symptoms. A score of 3 points is considered a cut-off point, in which further evaluation is recommended.
Patients' quality of life | within 1 week after patient assessment by the Enhanced Supportive Care Team
  Patients' quality of life assessed through the European Organisation for Research and Treatment of Cancer quality of life core 15 palliative questionnaire. This 15-item questionnaire, employs a 4-point Likert scale for each question, and the resulting scores are linearly transformed to a possible range of 0 to 100, where higher scores indicate a better quality of life
Trust in the treating oncologist | within 1 week after patient assessment by the Enhanced Supportive Care Team
  Patients' trust in the treating oncologist assessed on a numeric rating scale ranging from 0-10 with higher scores indicating more trust
Satisfaction with care | within 1 week after patient assessment by the Enhanced Supportive Care Team
  Patients' satisfaction with care assessed on a numeric rating scale ranging from 0-10 with higher scores indicating greater satisfaction

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Stone, Prof, Principal Investigator — University College, London; Joanna Sheppard, MD, Principal Investigator — University College London Hospital
Locations (1):
- University College Hospital Macmillan Cancer Centre, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bakitas MA, Tosteson TD, Li Z, Lyons KD, Hull JG, Li Z, Dionne-Odom JN, Frost J, Dragnev KH, Hegel MT, Azuero A, Ahles TA. Early Versus Delayed Initiation of Concurrent Palliative Oncology Care: Patient Outcomes in the ENABLE III Randomized Controlled Trial. J Clin Oncol. 2015 May 1;33(13):1438-45. doi: 10.1200/JCO.2014.58.6362. Epub 2015 Mar 23. PMID 25800768
- [Background] Bakitas M, Lyons KD, Hegel MT, Balan S, Brokaw FC, Seville J, Hull JG, Li Z, Tosteson TD, Byock IR, Ahles TA. Effects of a palliative care intervention on clinical outcomes in patients with advanced cancer: the Project ENABLE II randomized controlled trial. JAMA. 2009 Aug 19;302(7):741-9. doi: 10.1001/jama.2009.1198. PMID 19690306
- [Background] Chen CH, Kuo SC, Tang ST. Current status of accurate prognostic awareness in advanced/terminally ill cancer patients: Systematic review and meta-regression analysis. Palliat Med. 2017 May;31(5):406-418. doi: 10.1177/0269216316663976. Epub 2016 Aug 4. PMID 27492160
- [Background] El-Jawahri A, Traeger L, Park ER, Greer JA, Pirl WF, Lennes IT, Jackson VA, Gallagher ER, Temel JS. Associations among prognostic understanding, quality of life, and mood in patients with advanced cancer. Cancer. 2014 Jan 15;120(2):278-85. doi: 10.1002/cncr.28369. Epub 2013 Oct 10. PMID 24122784
- [Background] Enzinger AC, Zhang B, Schrag D, Prigerson HG. Outcomes of Prognostic Disclosure: Associations With Prognostic Understanding, Distress, and Relationship With Physician Among Patients With Advanced Cancer. J Clin Oncol. 2015 Nov 10;33(32):3809-16. doi: 10.1200/JCO.2015.61.9239. Epub 2015 Oct 5. PMID 26438121
- [Background] Epstein AS, Prigerson HG, O'Reilly EM, Maciejewski PK. Discussions of Life Expectancy and Changes in Illness Understanding in Patients With Advanced Cancer. J Clin Oncol. 2016 Jul 10;34(20):2398-403. doi: 10.1200/JCO.2015.63.6696. Epub 2016 May 23. PMID 27217454
- [Background] Fisher K, Seow H, Cohen J, Declercq A, Freeman S, Guthrie DM. Patient characteristics associated with prognostic awareness: a study of a Canadian palliative care population using the InterRAI palliative care instrument. J Pain Symptom Manage. 2015 Apr;49(4):716-25. doi: 10.1016/j.jpainsymman.2014.08.008. Epub 2014 Sep 8. PMID 25220047
- [Background] Glare PA, Sinclair CT. Palliative medicine review: prognostication. J Palliat Med. 2008 Jan-Feb;11(1):84-103. doi: 10.1089/jpm.2008.9992. PMID 18370898
- [Background] Greer JA, Pirl WF, Jackson VA, Muzikansky A, Lennes IT, Heist RS, Gallagher ER, Temel JS. Effect of early palliative care on chemotherapy use and end-of-life care in patients with metastatic non-small-cell lung cancer. J Clin Oncol. 2012 Feb 1;30(4):394-400. doi: 10.1200/JCO.2011.35.7996. Epub 2011 Dec 27. PMID 22203758
- [Background] Groenvold M, Petersen MA, Aaronson NK, Arraras JI, Blazeby JM, Bottomley A, Fayers PM, de Graeff A, Hammerlid E, Kaasa S, Sprangers MA, Bjorner JB; EORTC Quality of Life Group. The development of the EORTC QLQ-C15-PAL: a shortened questionnaire for cancer patients in palliative care. Eur J Cancer. 2006 Jan;42(1):55-64. doi: 10.1016/j.ejca.2005.06.022. Epub 2005 Sep 12. PMID 16162404
- [Background] Hausner D, Tricou C, Mathews J, Wadhwa D, Pope A, Swami N, Hannon B, Rodin G, Krzyzanowska MK, Le LW, Zimmermann C. Timing of Palliative Care Referral Before and After Evidence from Trials Supporting Early Palliative Care. Oncologist. 2021 Apr;26(4):332-340. doi: 10.1002/onco.13625. Epub 2021 Jan 2. PMID 33284483
- [Background] Hui D, Elsayem A, De la Cruz M, Berger A, Zhukovsky DS, Palla S, Evans A, Fadul N, Palmer JL, Bruera E. Availability and integration of palliative care at US cancer centers. JAMA. 2010 Mar 17;303(11):1054-61. doi: 10.1001/jama.2010.258. PMID 20233823
- [Background] Jackson VA, Jacobsen J, Greer JA, Pirl WF, Temel JS, Back AL. The cultivation of prognostic awareness through the provision of early palliative care in the ambulatory setting: a communication guide. J Palliat Med. 2013 Aug;16(8):894-900. doi: 10.1089/jpm.2012.0547. Epub 2013 Jun 20. PMID 23786425
- [Background] Janssens A, Derijcke S, Galdermans D, Daenen M, Surmont V, De Droogh E, Lefebure A, Saenen E, Vandenbroucke E, Morel AM, Sadowska A, van Meerbeeck JP. Prognostic Understanding and Quality of Life in Patients With Advanced Lung Cancer: A Multicenter Study. Clin Lung Cancer. 2019 May;20(3):e369-e375. doi: 10.1016/j.cllc.2018.11.011. Epub 2018 Dec 13. PMID 30635259
- [Background] Kennedy BM, Rehman M, Johnson WD, Magee MB, Leonard R, Katzmarzyk PT. Healthcare Providers versus Patients' Understanding of Health Beliefs and Values. Patient Exp J. 2017;4(3):29-37. PMID 29308429
- [Background] Kroenke K, Spitzer RL, Williams JB. The Patient Health Questionnaire-2: validity of a two-item depression screener. Med Care. 2003 Nov;41(11):1284-92. doi: 10.1097/01.MLR.0000093487.78664.3C. PMID 14583691
- [Background] Kuhne F, Hermann M, Preisler M, Rohrmoser A, Letsch A, Goerling U. Prognostic Awareness in Advanced Disease: A Review Update and Concept Analysis. Front Psychol. 2021 Jun 24;12:629050. doi: 10.3389/fpsyg.2021.629050. eCollection 2021. PMID 34248736
- [Background] Kurita K, Siegler EL, Reid MC, Maciejewski RC, Prigerson HG. It Is Not What You Think: Associations Between Perceived Cognitive and Physical Status and Prognostic Understanding in Patients With Advanced Cancer. J Pain Symptom Manage. 2018 Aug;56(2):259-263. doi: 10.1016/j.jpainsymman.2018.04.016. Epub 2018 May 10. PMID 29753102
- [Background] Li C, Friedman B, Conwell Y, Fiscella K. Validity of the Patient Health Questionnaire 2 (PHQ-2) in identifying major depression in older people. J Am Geriatr Soc. 2007 Apr;55(4):596-602. doi: 10.1111/j.1532-5415.2007.01103.x. PMID 17397440
- [Background] Mack JW, Fasciano KM, Block SD. Communication About Prognosis With Adolescent and Young Adult Patients With Cancer: Information Needs, Prognostic Awareness, and Outcomes of Disclosure. J Clin Oncol. 2018 Jun 20;36(18):1861-1867. doi: 10.1200/JCO.2018.78.2128. Epub 2018 Apr 23. PMID 29683788
- [Background] Mayer DK, Nasso SF, Earp JA. Defining cancer survivors, their needs, and perspectives on survivorship health care in the USA. Lancet Oncol. 2017 Jan;18(1):e11-e18. doi: 10.1016/S1470-2045(16)30573-3. PMID 28049573
- [Background] Sato T, Soejima K, Fujisawa D, Takeuchi M, Arai D, Nakachi I, Naoki K, Kawada I, Yasuda H, Ishioka K, Nukaga S, Kobayashi K, Masaki K, Inoue T, Hikima K, Nakamura M, Ohgino K, Oyamada Y, Funatsu Y, Terashima T, Miyao N, Sayama K, Saito F, Sakamaki F, Betsuyaku T. Prognostic Understanding at Diagnosis and Associated Factors in Patients with Advanced Lung Cancer and Their Caregivers. Oncologist. 2018 Oct;23(10):1218-1229. doi: 10.1634/theoncologist.2017-0329. Epub 2018 Aug 17. PMID 30120158
- [Background] Shen MJ, Trevino KM, Prigerson HG. The interactive effect of advanced cancer patient and caregiver prognostic understanding on patients' completion of Do Not Resuscitate orders. Psychooncology. 2018 Jul;27(7):1765-1771. doi: 10.1002/pon.4723. Epub 2018 Apr 30. PMID 29611241
- [Background] Shin JA, El-Jawahri A, Parkes A, Schleicher SM, Knight HP, Temel JS. Quality of Life, Mood, and Prognostic Understanding in Patients with Metastatic Breast Cancer. J Palliat Med. 2016 Aug;19(8):863-9. doi: 10.1089/jpm.2016.0027. Epub 2016 Apr 28. PMID 27124211
- [Background] Tang ST, Chang WC, Chen JS, Chou WC, Hsieh CH, Chen CH. Associations of prognostic awareness/acceptance with psychological distress, existential suffering, and quality of life in terminally ill cancer patients' last year of life. Psychooncology. 2016 Apr;25(4):455-62. doi: 10.1002/pon.3943. Epub 2015 Aug 17. PMID 26283000
- [Background] Tang ST, Wen FH, Hsieh CH, Chou WC, Chang WC, Chen JS, Chiang MC. Preferences for Life-Sustaining Treatments and Associations With Accurate Prognostic Awareness and Depressive Symptoms in Terminally Ill Cancer Patients' Last Year of Life. J Pain Symptom Manage. 2016 Jan;51(1):41-51.e1. doi: 10.1016/j.jpainsymman.2015.08.006. Epub 2015 Sep 18. PMID 26386187
- [Background] Thompson GN, Chochinov HM, Wilson KG, McPherson CJ, Chary S, O'Shea FM, Kuhl DR, Fainsinger RL, Gagnon PR, Macmillan KA. Prognostic acceptance and the well-being of patients receiving palliative care for cancer. J Clin Oncol. 2009 Dec 1;27(34):5757-62. doi: 10.1200/JCO.2009.22.9799. Epub 2009 Oct 13. PMID 19826116
- [Background] Zimmermann C, Swami N, Krzyzanowska M, Hannon B, Leighl N, Oza A, Moore M, Rydall A, Rodin G, Tannock I, Donner A, Lo C. Early palliative care for patients with advanced cancer: a cluster-randomised controlled trial. Lancet. 2014 May 17;383(9930):1721-30. doi: 10.1016/S0140-6736(13)62416-2. Epub 2014 Feb 19. PMID 24559581